CLINICAL TRIAL: NCT02418156
Title: A Post Market Observational Study on the Use of CorMatrix® ECM® for Femoral Arterial Reconstruction
Brief Title: A Study on the Use of CorMatrix® ECM® for Femoral Arterial Reconstruction
Acronym: PERFORM
Status: Completed | Type: Observational
Sponsor: Elutia Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-PR-1120
Record Dates: First submitted 2015-04-09; First posted 2015-04-16 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single Arm: Subjects undergoing femoral arterial reconstruction using CorMatrix ECM for vascular repair.
  Interventions: Device: CorMatrix ECM for Vascular Repair

INTERVENTIONS:
Device: CorMatrix ECM for Vascular Repair — Standard femoral arterial interventional procedure using CorMatrix ECM for vascular repair.

SUMMARY:
To gather information on the use of CorMatrix ECM for Vascular Repair in the reconstruction of the femoral artery.

DETAILED DESCRIPTION:
OBJECTIVE The objective of the study is to actively gather additional information on the use of CorMatrix ECM for vascular repair in the reconstruction of the femoral artery. The CorMatrix ECM for Vascular Repair may be used for patch closure of vessels, as a pledget, or for suture line buttressing when repairing peripheral vessels.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be undergoing femoral arterial reconstruction with patch angioplasty closure
2. Surgeon intends to use CorMatrix ECM per FDA cleared Indications for Use
3. Subject possesses ability to provide informed consent
4. Subject expresses understanding and willingness to fulfill all expected requirements of protocol

Exclusion Criteria:

1. Known sensitivity to porcine material

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting for femoral arterial reconstruction with patch angioplasty.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-05; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Observation of subjects undergoing femoral arterial reconstruction using CorMatrix ECM for vascular repair.
  CorMatrix ECM for Vascular Repair: Standard femoral arterial interventional procedure using CorMatrix ECM for arterial repair.
Period: Overall Study
Arm/Group | Single Arm
Started | 38
Completed | 21
Not Completed | 17
Not completed — Lost to Follow-up | 12
Not completed — Death | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Subject refused to return | 1

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Observation of subjects undergoing femoral arterial reconstruction using CorMatrix ECM for vascular repair.
  CorMatrix ECM for Vascular Repair: Standard femoral arterial interventional procedure using CorMatrix ECM for arterial repair.
  Device performance and adverse events were collected.
Arm/Group | Single Arm
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 15
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 38
Device Performance [Number; unit: Procedures] | 45
CoMorbidity Risk Factors [Number; unit: participants]
  Hypertension | 35
  Hyperlipidemia | 26
  Diabetes | 18
  Previous Vascular Surgery | 20
  Active tobacco use | 15
  Hx Sedentary lifestyle | 12
  Family Hx of Vascular Disease | 12
  Previous groin surgery | 13
  Hx of CABG | 10
  Previous MI | 9
  Hx of renal disease | 7
  Obesity | 3
Weight [Mean (Standard Deviation); unit: Pounds] | 177.3 (37.1)
Tobacco Use [Count of Participants; unit: Participants]
  Current smoker | 15
  Previous smoker | 18
  Never | 5
Indication for Surgery [Number; unit: Surgical Indications]
  Acute critical limb ischemia | 7
  Claudication (Fontaine class IIb) | 34
  Rest and night pain (Fontaine class III) | 4
  Gangrene (Fontaine class IV) | 2
  Infected prosthesis | 0
  Other | 2
Intervention/Procedure [Number; unit: Interventions/Procedures]
  Iliofemoral endarterectomy | 30
  Femoral endarterectomy | 11
  Iliofemoral endarterectomy with profundaplasty | 3
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Device-Related Adverse Events
Description: Proportion of patients experiencing device related adverse events.
Time Frame: Up to 12 months follow-up
Population: Several participants had both limbs treated resulting in a greater number of procedures than participants analyzed.
Measure: Number (95% Confidence Interval); unit: Proportion of Participants that Experien
Units Other Than Participants: Procedures
Arm/Group | Single Arm
Number analyzed (Participants) | 38
Number analyzed (Procedures) | 45
Proportion of Participants that Experien | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 2/38
Serious Adverse Events (participants affected / at risk) | 14/38
Other Adverse Events (participants affected / at risk) | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=38)
Depression and Suicide Attempt (Psychiatric disorders) | 1 (1)
Non Healing Lower Extremity Ulcer (Vascular disorders) | 1 (1)
Right upper lobe adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Failed Vascular Interventions/Severe PAD (Vascular disorders) | 1 (1)
Coag Neg Staph Bacteremia (Blood and lymphatic system disorders) | 1 (1)
Post Operative Seroma (Vascular disorders) | 1 (1)
Critical Limb Ischemia (Vascular disorders) | 1 (1)
Pseudoaneurysm (Surgical and medical procedures) | 1 (1) — Due to a broken suture along the medial line of anastomosis.
Stroke-like symptoms (Cardiac disorders) | 1 (1)
Atrial flutter & atrial fibrillation (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Bilaterial lower extremity pain and numbness (Vascular disorders) | 1 (1)
CVA (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT02418156/Prot_SAP_000.pdf